CLINICAL TRIAL: NCT04958980
Title: The Effectiveness of the Multiprofessional Approach in an Educational Group in the Control of Diabetes Mellitus in Patients Using Oral Hypoglycemic Agents From a Basic Health Unit in the City of Guarulhos/ SP: a Randomized Study
Brief Title: Multiprofessional Approach in Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leonardo Paroche de Matos (Other)
Responsible Party: Principal Investigator, Leonardo Paroche de Matos, main researcher, Leonardo Paroche de Matos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00129122020
Record Dates: First submitted 2020-12-29; First posted 2021-07-12 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus; Health education; Multiprofessional team; Collective health; Health promotion
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Health Education

STUDY DESIGN:
Intervention Model Description: randomized clinical study conducted in an educational group at the Basic Health Unit of Nova Bonsucesso with six monthly meetings scheduled with 24 patients with type II diabetes mellitus users of oral hypoglycemic agents divided into two subgroups: 12 users of the control group and 12 users of the study group (who will receive the researchers' interventions) and will be accompanied by laboratory tests and individual evaluations to verify the effectiveness of multiprofessional action in the control of diabetes mellitus.
Who Masked: Participant
Masking Description: The formation of randomized groups will occur by random drawing, obeying the proportion of 1: 1 in both groups, that is, 12 participants in each group (control and intervention) that will be selected after the screening carried out by the research nurse (to verify some possible exclusion criteria for research participants), reducing the occurrence of methodological bias in the sampling phase and ensuring the possibility that all participants can be included in the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (No Intervention): The control group will be evaluated in 2 stages: at the beginning and at the end of the study and will be accompanied only with scheduled medical consultations (also simulating the reality of basic health units with a traditional model of care) and the intervention group will undergo evaluations with the multiprofessional team on two occasions (at the beginning and at the end of the study)
- Specific and educational guidelines on pathology care (diabetes mellitus) (Active Comparator): Multiprofessional educational guidelines and analysis of the following exams:
  * Periodontal record, bleeding rate on and visible plaque;
  * Body mass index (BMI): weight (kg) divided by height squared (m²);
  * Serum glucose values;
  * Glycated hemoglobin;
  * Blood count: hemoglobin;
  * Urea: male:
  * Creatinine male;
  * Uric acid;
  * Oxalacetic glutamic transaminase;
  * Glutamic pyruvic transaminase;
  * Total cholesterol and fractions: Cholesterol, Non HDL, LDL, VLDL;
  * Triglycerides;
  * Type I urine;
  * Vitamin D3 25OH;
  * Microalbuminuria;
  * Blood pressure: systolic;
  * Abdominal circumference.
  Interventions: Behavioral: Specific and educational guidelines on care for pathology (diabetes mellitus) according to each profession involved in the research

INTERVENTIONS:
Behavioral: Specific and educational guidelines on care for pathology (diabetes mellitus) according to each profession involved in the research — Physician: Guidance on pathology, sequelae and treatment, as well as guidance on the importance of medical monitoring.
  Dental surgeon: guidance on oral health, demonstration of brushing techniques and daily flossing and periodontal changes resulting from diabetes mellitus.
  Nurse: Guidance on pathology prioritizing pathophysiology, self-care and skin care and wound prevention (vascular sequelae).
  Nutritionist: nutritional guidelines on diabetes mellitus and healthy eating habits.
  Physiotherapist: guidance on prevention of falls and injuries and health promotion.
  Physical educator: guidance on the importance of practicing physical activities for general health, encouraging self-care and body awareness and demonstrating basic physical activities that can be performed at home.
  Arms: Specific and educational guidelines on pathology care (diabetes mellitus)

SUMMARY:
OBJECTIVE: to verify the effectiveness of adopting the practice of educational groups in primary care and the multiprofessional role in the control of diabetes mellitus in adults. METHODOLOGY: a randomized clinical study carried out in an educational group at the Basic Health Unit Nova Bonsucesso with six monthly meetings scheduled with 24 patients with type II diabetes mellitus users of oral hypoglycemic agents divided into two subgroups: 12 users in the control group and 12 users in the control group. study (which will receive the interventions of the multidisciplinary team) and will be accompanied by laboratory tests and individual evaluations to verify the effectiveness of the multidisciplinary action in the control of diabetes mellitus.

DETAILED DESCRIPTION:
INTRODUCTION: diabetes mellitus is highlighted as an obstacle in health equipment because it is a chronic disease and has a high mortality rate. The pathology results in hyperglycemia, disorders or insufficiency of several organs. OBJECTIVE: to verify the effectiveness of adopting the practice of educational groups in primary care and the multidisciplinary role in the control of diabetes mellitus in adults. THEORETICAL BACKGROUND: type II diabetes mellitus (type II DM) is a pathology that represents a high risk for cardiovascular, renal, ophthalmological complications and in several other systems. It is considered a major issue to be controlled by health services, as the high cost of treatments related to the sequelae of type II DM, as well as high rates of hospitalizations and associated therapies have been increasing and decompensating public budgets. Primary care has a fundamental role in preventing the disease and associated complications. METHODOLOGY: randomized clinical study conducted in an educational group at the Basic Health Unit Nova Bonsucesso with six monthly meetings scheduled with 24 patients with type II diabetes mellitus users of oral hypoglycemic agents divided into two subgroups: 12 users in the control group and 12 users in the group study (which will receive the interventions of the multidisciplinary team) and will be accompanied by laboratory tests and individual evaluations to verify the effectiveness of the multidisciplinary performance in the control of diabetes mellitus. RESULTS: the participants are expected to show improvements in the control of the pathology and awareness about the relevance of self-care, facts that will be observed through laboratory data and subsequent multi-professional evaluations.

ELIGIBILITY:
Inclusion Criteria:

* 24 on-insulin-dependent type II diabetes patients (users of oral hypoglycemic agents),
* over 18 years of age,
* both sexes,
* with no restrictions on physical exercise (found after medical evaluation)
* who agreed to participate voluntarily in the study (after signature of the Free and Informed Consent Form)
* of a specific area of the Family Health Strategy - chosen by the proximity to the Basic Health Unit.

Exclusion Criteria:

* Patients with associated pathologies: cardiovascular conditions: Congestive Heart Failure,Decompensated Systemic Arterial Hypertension, Sequela of Acute Myocardial Infarction
* Cancer patients,
* Respiratory conditions: Chronic Obstructive Pulmonary Disease, Severe asthma and any other disabling lung condition.
* Endocrine conditions that aggravate diabetes mellitus: Pancreatic pathologies (pancreatitis, pancreatic cysts, obstructions and pancreatic cancer)
* Patients with impaired vision,
* Motor or balance disorders,
* With any special needs (physical or intellectual),
* With consequences resulting from the evolution of type II diabetes mellitus
* Users who refused to participate in the research.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
incidence of periodontitis associated with diabetes mellitus | 6 months
  Periodontal record: up to 3mm.
Risk rate for periodontal disease (in %) associated with diabetes mellitus | 6 months
  Bleeding rate on and visible plaque: up to 10%;
Association of glycemic control with changes in body weight (in kg) | 6 months
  Body mass index (BMI): weight (kg) divided by height squared (m²);
Comparison of glycemic control | 6 months
  Serum glucose values: 80 to 130mg/ dl
% of participants at risk for worsening diabetes mellitus | 6 months
  Glycated hemoglobin: <7%
% of participants at risk for anemic diseases | 6 months
  Blood count: hemoglobin: male 13-17g/ dl, female: 12 -15g/ dl
Concentration of participants at risk for developing kidney complications [urea] | 6 months
  Urea: male: <40mg/ dl, female: <55mg/ dl
Concentration of participants at risk of developing kidney failure | 6 months
  Creatinine male: 0.7-1.30mg/ dl, female: 0.5- 1.10mg/ dl
Concentration of participants at risk for the development of kidney stones and worsening of diabetes mellitus | 6 months
  Uric acid: male: 3.4- 7.0mg/ dl, female: 2.4- 7.4mg/ dl
Concentration of participants at risk for the development of liver complications | 6 months
  Oxalacetic glutamic transaminase: male: <50U/ L, female: <40U/ L
Concentration of participants at risk for the development of liver failure associated with diabetes mellitus | 6 months
  Glutamic pyruvic transaminase: male: <50U/ L, female: <40U/ L
Observation of the risk of developing cardiovascular diseases associated with diabetes mellitus | 6 months
  Total cholesterol and fractions: Cholesterol: 190mg/ dl, HDL:> 40mg/ dl, Non HDL: <160mg/ dl, LDL: <100mg/ dl, VLDL: 10- 50mg/ dl
Observation of triglyceride rates and the development of risk for cardiovascular complications associated with diabetes mellitus | 6 months
  Triglycerides: <175mg/ dl
Concentration of participants with renal complications and urinary glucose and protein elimination associated with diabetes mellitus | 6 months
  Type I urine: negative proteinuria and glycosuria
Concentration of participants at increased risk for diabetes complications related to vitamin D deficiency | 6 months
  Vitamin D3 25OH: <60y: >20ng/ dl, >60y: >30ng/dl
Observation of the risk of developing nephropathies, retinopathies and cardiovascular diseases associated with diabetes mellitus | 6 months
  Microalbuminuria: <30mg/day
Concentration of participants at risk of developing systemic arterial hypertension associated with diabetes mellitus | 6 months
  Blood pressure: systolic- <130mmHg, diastolic: <85mHg
Concentration of participants at increased risk for diabetes complications related to increased waist circumference | 6 months
  Abdominal circumference: male: 102cm, female: 88cm

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Oliveira, Principal Investigator — Guarulhos City Hall

IPD SHARING:
Plan to Share IPD: No